CLINICAL TRIAL: NCT01235364
Title: Assessment of Pain With Insertion of the Foley Catheter for Induction of Labour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Dr. Maria Jonsson, Department of obstetrics and gynecology, Uppsala University Hospital. Uppsala
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-nr 2009/ 218
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Pain
Keywords: Foley catheter; induction; labour; skin conductance; visual analogue scale; mechanical method
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Digital (Experimental): The patient was randomized to digital insertion of the Foley catheter
  Interventions: Device: Foley catheter
- Speculum (Experimental)
  Interventions: Device: Foley catheter

INTERVENTIONS:
Device: Foley catheter — The Foley catheter was placed with the digital method
  Arms: Digital
Device: Foley catheter — The Foley catheter was placed with a speculum
  Arms: Speculum

SUMMARY:
The purpose of this study is to assess pain in women randomised to digital or speculum placement of a Foley catheter. Pain during cervical ripening with the Foley catheter is also to be evaluated as well as maternal satisfaction with induction of labour.

DETAILED DESCRIPTION:
The most common method described for placing the Foley catheter is under direct visualisation of the cervix during a sterile speculum examination. Another method is to place the catheter during a digital cervical examination.

Maternal discomfort/pain during speculum placement of the catheter has been evaluated in a few studies whereas studies that compare the digital method with the speculum method of placement are lacking.

The visual analogue scale is used to subjectively assess pain. With a skin conductance algesimeter an objective assessment of pain is possible.

ELIGIBILITY:
Inclusion Criteria:

* singleton fetus in cephalic presentation with a Bishop score of 3-5 and
* indication for induction of labour

Exclusion Criteria:

* low-lying placenta,
* undiagnosed vaginal bleeding,
* more than one previous caesarean section,
* previous use of an induction or pre-induction agent during the same pregnancy,
* signs of infection (maternal fever)
* non- proficiency in the Swedish language.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Pain assessed by VAS and SCA, in women randomised to digital or speculum placement of a Foley catheter. | At insertion of Foley catheter

SECONDARY OUTCOMES:
To assess pain with VAS and SCA during cervical ripening with the Foley catheter and to evaluate maternal satisfaction. To evaluate if markers of stress in blood and amniotic fluid correlate with VAS and SCA. | During treatment with Foley catheter. At expulsion of Foley catehter

CONTACTS AND LOCATIONS:
Locations (1):
- Department of obstetrics and gynecology, Uppsala university hospital, Uppsala, Sweden